CLINICAL TRIAL: NCT00348803
Title: Gene Mutations in Secondary Pulmonary Hypertension
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Other Study IDs: 01
Record Dates: First submitted 2006-07-05; First posted 2006-07-06 (Estimated); Last update posted 2006-07-06 (Estimated); Status verified 2006-06

CONDITIONS: Chronic Thromboembolic Pulmonary Hypertension

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

SUMMARY:
As a pulmonary hypertension center, we have created a database that prospectively tracks patients with different forms of secondary pulmonary hypertension. Records include genetic analysis, and clinical and hemodynamic profiles.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CTEPH and patient consent

Exclusion Criteria:

* No patient consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Irene Lang, MD, Principal Investigator — Medical University of Vienna
Locations (1):
- Medical University of Vienna, Vienna, Austria